CLINICAL TRIAL: NCT01230047
Title: Evaluation of a Psychoeducational Intervention Teaching Mindfulness and Lifestyle Interventions for Clinical Depression and Anxiety (A Pilot Study)
Brief Title: Mindfulness and Lifestyle Interventions for Depression and Anxiety: A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arizona State University (Other)
Responsible Party: Jeffrey R. Lacasse, College of Public Programs, Arizona State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1018
Record Dates: First submitted 2010-10-19; First posted 2010-10-28 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-10

CONDITIONS: Depression; Anxiety; Major Depression
Keywords: depression; anxiety; psychoeducation; self-help; psychosocial
MeSH Terms: conditions — Depression; Anxiety Disorders; Depressive Disorder, Major | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychoeducational Course (Experimental): In this arm, clients receive the psychoeducational course.
  Interventions: Behavioral: Psychoeducational course
- Treatment-as-usual/Waiting list (No Intervention): Clients assigned to this condition will receive treatment-as-usual (TAU) and be placed on a waiting list.

INTERVENTIONS:
Behavioral: Psychoeducational course — Psychoeducational course on mindfulness and lifestyle interventions for depression and anxiety
  Other Names: Psychoeducational, therapeutic, psychosocial, self-help
  Arms: Psychoeducational Course

SUMMARY:
This is a quasi-experimental evaluation of psychoeducational course focusing on mindfulness and lifestyle changes for depression and anxiety; clients in active treatment group are compared to those in a treatment-as-usual wait-list control group. The primary hypothesis is that the psychoeducational course will result in lower levels of depression and anxiety as compared to the wait-listed treatment-as-usual comparison group.

DETAILED DESCRIPTION:
This study evaluates a psychoeducational intervention: Teaching mindfulness and lifestyle interventions to adult clients who self-report problems with depression and/or anxiety. The course is eight weeks long. Clients are assigned to either (1) receive the course (COU condition) from October- December 2010 or (2) placed on a waiting list and receive treatment-as-usual (TAU condition). Those in the TAU group will be offered the course in January 2011.

Random assignment to COU or TAU conditions will be attempted although this may be relaxed due to institutional constraints.

Participants are assessed on the Beck Depression Inventory (BDI) and Beck Anxiety Inventory (BAI) at the beginning of the course, on the last day of the course, at 1-month post-course, at 4-months post-course, and at 12-months post-course.

Participants in the COU condition will be compared to those in TAU condition at the beginning of the course, on the last day of the course, and at 1-month post-course. Further evaluations (4 and 12 months post-course) will be pre-post evaluations without a comparison group.

ELIGIBILITY:
Inclusion Criteria:

* Participants self-report as having depression or anxiety
* Adults (age 18 or above)
* Clients willing to participate in an 8-week psychoeducational course

Exclusion Criteria:

* A diagnosis of a psychotic disorder
* Unwilling to participate in 8-week psychoeducational course

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-01 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory (BDI) | BDI administered at 12 weeks
  Depression will be assessed by comparing BDI scores on day one with BDI scores at twelve weeks (four weeks after conclusion of the psychoeducational course).
  The primary study hypothesis is that the psychoeducational course group will have a greater reduction in BDI scores when compared to the treatment-as-usual wait-listed comparison group.

SECONDARY OUTCOMES:
Beck Anxiety Inventory (BAI) | BAI administered at 8 weeks
Beck Anxiety Inventory (BAI) | BAI administered at 12 weeks
Beck Anxiety Inventory (BAI) | BAI administered at 24 weeks
Beck Anxiety Inventory (BAI) | BAI administered at 60 weeks
Beck Depression Inventory (BDI) | BDI administered at 8 weeks
Beck Depression Inventory (BDI) | BDI administered at 24 weeks
Beck Depression Inventory (BDI) | BDI administered at 60 weeks
Beck Anxiety Inventory (BAI) | BAI administered at Day 1 of Study
Beck Depression Inventory (BDI) | BDI administered at Day 1 of Study
Client Medication Use | Measured on Day 1 of Study
  Clients fill out a survey which includes a question asking if they are currently taking psychiatric medication.
Client Medication Use | Measured at 8 weeks
  Clients fill out a survey which includes a question asking if they are currently taking psychiatric medication.
Client Medication Use | Measured at 12 weeks
  Clients fill out a survey which includes a question asking if they are currently taking psychiatric medication.
Client Medication Use | Measured at 24 weeks
  Clients fill out a survey which includes a question asking if they are currently taking psychiatric medication.
Client Medication Use | Measured at 60 weeks
  Clients fill out a survey which includes a question asking if they are currently taking psychiatric medication.
Client Currently Seeing Therapist | Measured on Day 1 of study
  Clients are given a survey which includes a question asking if they are currently seeing a clinician for psychotherapy.
Client Currently Seeing Therapist | Measured at week 8
  Clients are given a survey which includes a question asking if they are currently seeing a clinician for psychotherapy.
Client Currently Seeing Therapist | Measured at week 12
  Clients are given a survey which includes a question asking if they are currently seeing a clinician for psychotherapy.
Client Currently Seeing Therapist | Measured at week 24
  Clients are given a survey which includes a question asking if they are currently seeing a clinician for psychotherapy.
Client Currently Seeing Therapist | Measured at week 60
  Clients are given a survey which includes a question asking if they are currently seeing a clinician for psychotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Lacasse, PhD, Principal Investigator — Arizona State University
Locations (1):
- Utah Youth Village, Salt Lake City, Utah, United States